CLINICAL TRIAL: NCT00862472
Title: Safety and Efficacy Study of DuoTrav APS Versus DuoTrav
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Management decision not to conduct an additional efficacy study.
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-006
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: open-angle glaucoma; ocular hypertension; open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component)
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Duotrav

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DuoTrav APS (Experimental): DuoTrav APS QD AM
  Interventions: Drug: DuoTrav APS
- DuoTrav (Active Comparator): DuoTrav QD AM
  Interventions: Drug: DuoTrav

INTERVENTIONS:
Drug: DuoTrav APS — DuoTrav APS QD AM
  Arms: DuoTrav APS
Drug: DuoTrav — DuoTrav QD AM
  Arms: DuoTrav

SUMMARY:
The purpose of the study is to demonstrate that the IOP-lowering efficacy of DuoTrav APS, dosed once-daily in the morning, is non-inferior to that of DuoTrav, dosed once-daily in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with open-angle glaucoma or ocular hypertension who would benefit from a fixed combination medication, in the opinion of the investigator and who are currently on a stable treatment of IOP-lowering medication

Exclusion Criteria:

* VA not worse than 0.60
* additional clinically relevant ocular or systemic conditions may be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure (IOP) | 3 Months